CLINICAL TRIAL: NCT05545566
Title: Evaluation of Thoracic Ultrasound in Monitoring Pleural Drainage in Postoperative Thoracic Surgery
Acronym: EchTHor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 87RI22_0022 (EchTHor)
Record Dates: First submitted 2022-09-10; First posted 2022-09-19 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Thoracic Ultrasound; Pleural Drain Removal
Keywords: postoperative thoracic surgery; discharge decision; thoracic ultrasound; pleural drain removal; chest X-ray; thoracic surgery monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental)
  Interventions: Procedure: Thoracic ultrasound versus chest X-ray

INTERVENTIONS:
Procedure: Thoracic ultrasound versus chest X-ray — Perform un ultrasound test, in addition to Chest X-Ray (usual practice), few hours after the surgery (D0), the next day (D1) and 4 to 6 hours after drain removal.
  The data are collected in the standardized protocol for the two type of imaging.
  The thoracic ultrasound and the Chest X-Ray are performed, blindly each other, in the same position for the patient and the same suction level of drain.

SUMMARY:
The investigator would like to conduct a study in patients undergoing thoracic surgery to evaluate the effectiveness of thoracic ultrasound in the decision to discharge the patient after pleural drain removal.

DETAILED DESCRIPTION:
Thoracic drainage is a common and almost systematic practice after thoracic surgery requiring daily management and monitoring until and after its removal.

It allows, after opening the pleura, the evacuation of liquid and/or air retained in the pleural cavity.

The overall monitoring of the patient after thoracic surgery is based on clinical vigilance combined with thoracic imaging, in particular the chest X-ray which remains the Gold Standard (reference examination).

The removal of the drain is decided according to the quantity and appearance of the evacuated fluid, the persistence of air leaks, etc… A few hours after the removal of the drain, it is routine to perform a chest X-ray before authorizing a possible discharge from the department.

This practice does not correspond to an established scientific protocol but is systematically performed in our department before discharge.

Several studies have defended the place of ultrasound in thoracic imaging and its contribution to the detection of postoperative and intensive care complications.

Unlike radiography, this technique is non-irradiating, less expensive and more readily available. It allows the detection of pneumothorax, pleural effusions and other complications detectable on X-ray.

To our knowledge, the contribution of thoracic ultrasound has not been studied in the decision to authorize the discharge of the patient after removal of the thoracic drain.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing thoracic surgery (lung resection, pleural symphysis, biopsy or resection of a mediastinal tumor or ganglion, pleural decortication/decalcification) admitted immediately after surgery in the thoracic surgery department (standard care or continuous care) of the University Hospital of Limoges.

Exclusion Criteria:

* Admission to the intensive care unit after thoracic surgery.
* Pneumonectomy
* Chest wall surgery
* Patients <18 years old
* Not affiliated to social security
* Under guardianship or curatorship
* Pregnant women
* Not knowing the French language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Theoretical patient discharge | At the study completion, an average of 10 days
  Theoretical patient discharge based on imaging data (pleural ultrasound or chest x-ray):
  * YES: Score ≤ 2 on each of the 4 items assessed AND total score ≤ 4.
  * NO: Score ≥ 3 on each of the items assessed and/or total score ≥ 5.

SECONDARY OUTCOMES:
Pain du to examination | Day 0, Day 1 and At the study completion, an average of 10 days
  To compare the pain generated by each examination (thoracic radiography and pleural ultrasound) with Visual Analogic Scale (0 to 10) at Day 0, Day 1 and post-drainage)
Subcutaneous emphysema | Day 0, Day 1 and At the study completion, an average of 10 days
  Evaluation of the concordance of pleural ultrasound data and chest radiography on the presence of subcutaneous emphysema at D0, D1 and post drain removal.
Pneumothorax | Day 0, Day 1 and At the study completion, an average of 10 days
  Evaluation of the concordance of pleural ultrasound data and chest radiography on the presence of Pneumothorax at D0, D1 and post drain removal.
Pleural effusion | Day 0, Day 1 and At the study completion, an average of 10 days
  Evaluation of the concordance of pleural ultrasound data and chest radiography on the presence of Pleural effusion at D0, D1 and post drain removal.
Pulmonary Condensation | Day 0, Day 1 and At the study completion, an average of 10 days
  Evaluation of the concordance of pleural ultrasound data and chest radiography on the presence of Pulmonary Condensation at D0, D1 and post drain removal.

CONTACTS AND LOCATIONS:
Locations (1):
- Limoges Univesity Hospital, Limoges, France

IPD SHARING:
Plan to Share IPD: No